CLINICAL TRIAL: NCT00429546
Title: Maternal HIV: Intervention to Assist Disclosure to Children
Brief Title: Assisting HIV-infected Mothers in Disclosing Their Serostatus to Their Children
Acronym: TRACK
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Debra A. Murphy, Ph.D., Professor in Residence, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: R01MH077493 (NIH); R01MH077493 (NIH); DAHBR 9A-ASAP
Record Dates: First submitted 2007-01-29; First posted 2007-01-31 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2013-06

CONDITIONS: HIV
Keywords: Disclosure; Serostatus
MeSH Terms: interventions — Educational Status; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Participants will receive a cognitive-behavioral intervention designed to improve mother-child communication and parenting skills and prepare caregiver for disclosure of HIV serostatus to child
  Interventions: Behavioral: Teaching, Raising, and Communicating with Kids (TRACK)
- Control (Active Comparator): Participants will receive treatment as usual
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Teaching, Raising, and Communicating with Kids (TRACK) — TRACK is cognitive-behavioral treatment designed to improve mother-child communication and parenting skills and prepare caregiver for disclosure of HIV serostatus to child. The treatment consists of three 75-minute sessions that focus on exploring mothers' concerns, determining children's readiness to receive the news, planning for disclosure, and practicing disclosure.
  Arms: Intervention
Other: Treatment as usual — Treatment as usual includes standard care for HIV infected mothers.
  Arms: Control

SUMMARY:
This study will develop and evaluate the effectiveness of an intervention designed to assist HIV-infected mothers of young children in determining whether and how to appropriately disclose their HIV serostatus to their children.

DETAILED DESCRIPTION:
HIV is a serious, life threatening illness that requires a lifetime of treatment and disease management. Studies have shown that it can be very difficult for infected mothers to decide whether and/or when to disclose their HIV serostatus to their uninfected children. HIV-infected parents struggle with the fear that their children will be forced to grow up too quickly, become worried or depressed, or be angry with their parents once they learn that their parents have HIV. Family-based intervention programs have been successful in helping facilitate the disclosure process. This study will develop and evaluate the effectiveness of an intervention designed to assist HIV-infected mothers of young children in determining whether and how to appropriately disclose their HIV serostatus to their children.

Participants in this study will be randomly assigned to either the intervention or a standard of care condition. The intervention will consist of three 75-minute sessions that will focus on exploring mothers' concerns, determining children's readiness to receive the news, planning for disclosure, and practicing disclosure. Participants will also receive one follow-up phone call from the therapist about 3 weeks after the last session. Sessions will be scheduled at times that are convenient for the participants and therapists. Follow-up visits will include both mothers and their children, and will be held at Months 3, 6, and 9 following the end of the intervention. Assessments will include readiness to disclose HIV serostatus, mental health indicators, and family functioning.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of mother's HIV/AIDS status
* Healthy child (i.e., HIV uninfected) who is between 6 and 12 years of age and is unaware of maternal serostatus
* Mother is primary caregiver and child resides with her
* English- or Spanish-speaking

Exclusion Criteria:

* Child does not meet screening criteria (e.g., diagnosed with depression or suicide attempt, IQ score less than 75)
* Psychosis of parent or child (as advised by recruitment site clinicians)
* Child refuses to give assent

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2007-09; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Readiness to disclose HIV serostatus | Measured at Months 3, 6, and 9
Disclosure of HIV serostatus | Measured at Months 3, 6, and 9

SECONDARY OUTCOMES:
Mothers' mental health indicators | Measured at Months 3, 6, and 9
Children's mental health indicators | Measured at Months 3, 6, and 9
Children's behavioral problems | Measured at Months 3, 6, and 9
Parent-child relationship and family functioning | Measured at Months 3, 6, and 9

CONTACTS AND LOCATIONS:
Overall Officials: Debra A. Murphy, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States